CLINICAL TRIAL: NCT01273259
Title: Study of Dehydroepiandrosterone (DHEA) in Respiratory Pulmonary Hypertension in Adults. Phase 2 Trial
Brief Title: Study of Dehydroepiandrosterone (DHEA) in Respiratory Pulmonary Hypertension in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2003/04
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypertension, Pulmonary
Keywords: Hypertension, pulmonary; DHEA; six-minute walk test; pulmonary arterial pressure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 200 mg /day arm (Experimental)
  Interventions: Drug: DHEA Treatment
- 25 mg/day arm (Experimental)
  Interventions: Drug: DHEA Treatment

INTERVENTIONS:
Drug: DHEA Treatment — DHEA : 200 mg/day hard gelatine capsule
  Arms: 200 mg /day arm
Drug: DHEA Treatment — DHEA : 25 mg/day hard gelatine capsule
  Arms: 25 mg/day arm

SUMMARY:
DHEA prevents and reverses chronic hypoxic pulmonary hypertension in a chronic hypoxic-pulmonary hypertension model in the rat. However, no study has been performed in human. The purpose of this study is to determine if DHEA is effective in the treatment of respiratory pulmonary hypertension in adults with Chronic Obstructive Pulmonary Disease (COPD) on exercise capacity and haemodynamic variables. Patients will receive after randomisation either 25 mg/day or 200mg/day oral DHEA over a one-year period. Evaluation concerns clinical parameters, echocardiography and right catheterization after and before treatment. Primary end-point is the six-minute walk test. This is a prospective double blind, randomised, placebo controlled study which will be realized in four university hospitals in France : Bordeaux, Strasbourg, Toulouse and Limoges.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years old
* Chronic Obstructive Pulmonary Disease with FEVs/VC < 70% (*)
* Respiratory pulmonary hypertension with mean pulmonary arterial pressure ≥ 20 mmHg (*) related to normal pulmonary capillar pressure assessed by catheterization of the right side of the heart (pulmonary capillary wedge pressure ≤12mmHg)
* PO2 ≤ 70 mmHg assessed by arterial gasometry at ease
* If oxygenotherapy then oxygenotherapy more than 6 months before pre-screening
* Written informed consent

(*) Criteria assessed from last health check or the last exams for COPD diagnosis

Exclusion Criteria:

* clinical instability and/or respiratory exacerbation dangerous for catheterization
* Pregnancy (ßHCG > 20 UI /l) or breastfeeding on going
* General corticotherapy > 0,5 mg/kg/day prednisolon equivalent
* Hepatic insufficiency (TP < 50%) or renal insufficiency (creatininemia > 130 µmol/l) or diabetes mellitus type I or II (treated by oral antidiabetic or insulin)
* Left-heart failure (coronary heart disease and/or left valvulopathy)
* High level of prostatic specific antigen (PSA) (> 7ng/ml)
* Cancer antecedent or treatment on going

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05-06 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2015-06-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of DHEA on exercise capacity (six-minute walk test) | inclusion and one year of treatment

SECONDARY OUTCOMES:
Pulmonary and systemic arterial pressures (mean, systolic and diastolic) | Inclusion and after one year of treatment
Pulmonary vascular resistances | Inclusion and after one year of treatment
Safety / Compliance | along one year of treatment

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - University Hospital, Bordeaux, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse